CLINICAL TRIAL: NCT00441532
Title: A Double-Blind Randomized Study On Lidocaine Vs. Placebo Pain Control During Transrectal Ultrasound Guided Prostate Biopsy
Brief Title: Study On Lidocaine Vs. Placebo Pain Control During Transrectal Ultrasound Guided Prostate Biopsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Corewell Health East (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2005-117
Record Dates: First submitted 2007-02-28; First posted 2007-03-01 (Estimated); Last update posted 2011-11-23 (Estimated); Status verified 2010-10

CONDITIONS: Prostate Cancer
Keywords: prostate
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Lidocaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Lidocaine

SUMMARY:
Patients at risk for having prostate cancer usually undergo a biopsy of their prostate. This is most often done in the private urology office. Recent studies have suggested that injection of local anesthesia (lidocaine) near the nerves of the prostate will improve pain sensation during the biopsy procedure. Local anesthesia can be given through a separate needle through the rectal probe just prior to biopsy. However, many urologists to date perform their biopsies without anesthesia. Some claim that the needle used for anesthesia causes pain itself. Others claim that the pain is so minimal that the additional use of lidocaine (and extra time) is not necessary. We plan to reexamine the use of lidocaine and perform the first study where each patient will receive lidocaine and placebo on separate sides of their prostate.

DETAILED DESCRIPTION:
Patients at risk for having prostate cancer usually undergo a biopsy of their prostate. This is most often done in the private urology office. A probe with an ultrasound is inserted into the rectum of the patient and biopsies are taken with a spring-loaded needle. Most urologists take four to six biopsies of each side of the prostate. Years ago, biopsies were traditionally done without any anesthesia. Patients experienced some pain with each firing of the spring-loaded needle, but this is generally tolerable. Recent studies have suggested that injection of local anesthesia (lidocaine) near the nerves of the prostate will improve pain sensation during the biopsy procedure. Local anesthesia can be given through a separate needle through the rectal probe just prior to biopsy. However, many urologists to date perform their biopsies without anesthesia. Some claim that the needle used for anesthesia causes pain itself. Others claim that the pain is so minimal that the additional use of lidocaine (and extra time) is not necessary. We plan to reexamine the use of lidocaine and perform the first study where each patient will receive lidocaine and placebo on separate sides of their prostate.

Patients will undergo the traditional prostate biopsy procedure. They will be in the urology center at William Beaumont Hospital. Patients will lie on their side and an ultrasound probe will be inserted into the rectum. The size of the prostate will be measured with the ultrasound probe. A study coordinator will hand the physician a syringe containing either 2.5mL of lidocaine or saline (placebo). Neither the patient nor the physician will know which solution the syringe contains. The 2.5mL of the first syringe will be injected in the traditional area that local anesthesia is injected (periprostatic area) on the right side. Next, the second syringe will be handed to the physician containing the opposite drug (lidocaine or saline) and the physician will inject this on the left side. Four to six biopsies will be taken on the right side, and the study coordinator will record patient pain on a 1 to 10 scale after injection of the 2.5mL, and after each biopsy. Biopsies will then be taken on the left side, and again, study coordinators will record results of patient pain on a 1 to 10 scale. At the end of the procedure, patients will be given a questionnaire to assess overall pain, tolerability of the procedure, and whether or not they could tell which side of their prostate received the anesthesia.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are undergoing prostate ultrasound-guided biopsy from the practice of Drs. Diokno and Hollander.
2. Patients must speak English.
3. Patients must sign consent form.

Exclusion Criteria:

1. Patients having received prior radiation to the pelvic area.
2. Patients with any neurologic disorder that may interfere with pain sensation during biopsy.
3. Allergy to Lidocaine
4. Patients requiring additional anesthesia (e.g. anxiolytics)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2005-08; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
To determine if patients experience a significant difference in pain on the side of their prostate that had local anesthesia.

SECONDARY OUTCOMES:
To determine if patients feel that they could tolerate such a procedure with no anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Ananias Diokno, M.D., Principal Investigator — Corewell Health East
Locations (1):
- William Beaumont Hospital, Royal Oak, Michigan, United States